CLINICAL TRIAL: NCT03587571
Title: Prospective, Randomized Multi-center Study Comparing Function, Pain and Return to Work in Conservative Versus Surgical Treated Stable Lateral Malleolar Fractures
Brief Title: Comparing Function, Pain and Return to Work in Conservative Versus Surgical Treated Stable Lateral Malleolar Fractures
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient patient recruitment
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-01041
Record Dates: First submitted 2018-06-28; First posted 2018-07-16 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Malleolus Fracture, Lateral
MeSH Terms: conditions — Ankle Fractures | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Comparison of two established treatment options. Prospective, randomised (central block randomisation) multi-center clinical trial.
  The two treatment options (operative versus conservative) are split in two study arms and compared to each other. Patients are randomly allocated to one of the two study arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical intervention (Active Comparator): Open reduction and osteosynthesis by plating is done. Further after treatment is similar to conservative treatment arm.
  Interventions: Procedure: Surgical intervention
- Conservative treatment (No Intervention): At the first visit a split cast is applied. Afterwards physiotherapy and weightbearing as tolerated is allowed.

INTERVENTIONS:
Procedure: Surgical intervention — Open reduction and plate osteosynthesis.
  Arms: Surgical intervention

SUMMARY:
Ankle fractures are one of the most common fractures in adults resulting in hospital stays and inability to work. Instable or dislocated ankle fractures are mostly treated by surgery. Treatment of stable lateral ankle fractures is still discussed controversial. They can be treated conservatively as well as by surgery.

Furthermore, optimal aftercare is part of on-going discussion in both groups. Goal of any treatment is a fast, good functional outcome with pain free patients at low overall costs. Long-term results in terms of osteoarthritis should be kept in mind.

The investigators seek to compare conservative and operative treatment in stable lateral ankle fractures in a prospective, randomised trial.

The hypothesis is that there is no difference between conservative and surgically treated stable lateral malleolar fractures regarding pain, function, and return to the workplace.

DETAILED DESCRIPTION:
Ankle fractures are one of the most common fractures in adults resulting in hospital stays and inability to work. Instable or dislocated ankle fractures are mostly treated by surgery. Treatment of stable lateral ankle fractures is still discussed controversial. They can be treated conservatively as well as by surgery.

Furthermore, optimal aftercare is part of on-going discussion in both groups. Goal of any treatment is a fast, good functional outcome with pain free patients at low overall costs. Long-term results in terms of osteoarthritis should be kept in mind.

Primary study objective is the comparison of functional result after conservative versus operative treatment in stable lateral ankle fractures.

Secondary study objectives are the return to work, pain, and osteoarthritis. It is a prospective, randomised (site stratified block randomisation) multi-center clinical trial. The two treatment options are split in two study arms and compared to each other.

Measurements and procedures:

People with acute stable lateral malleolar fracture type Weber B are potential participants. Patients are recruited at their first visit in the emergency department or on the first contact with the orthopaedic department. They have to live in Switzerland in order to be able to show up at the regular visits. They have to work in order to gain information concerning the timeframe for return to work.

No vulnerable participants are included. The two treatment options (operative versus conservative) are split in two study arms and compared to each other. Patients are randomly allocated to one of the two study arms. A central block randomisation with 80 participants per block is installed in REDCap. At time of participating in the study, REDCap is assigning the patient to one of the study groups.

After enrolling in the study at the first visit a split cast is applied in both group. Surgical intervention should be performed within 2 weeks after trauma. The exact time of surgery is determined by the treating surgeon and documented. In the surgical group open reduction and osteosynthesis by plating is done.

In the conservative group clinical and radiological re-evaluation is done within the first 2 weeks after trauma.

Both groups are further treated with an orthosis and allowed to bear weight as possible.

At time of accident, within the first two weeks, after 6 and 12 weeks, after 1, 3 and 5 years the patient is examined clinically and radiologically. Olerud Molander Ankle Score (OMAS), Foot Function Index (FFI), American Orthopaedic Foot and Ankle Society Score (AOFAS), Visual Analogue Scale Foot and Ankle (VAS FA) and epidemiological and clinical findings are gathered. Patients who do not reach the 12 weeks follow-up will be considered drop-outs and must be replaced. In accordance to the intention to treat analysis (ITT-analysis) data will be included in the statistical analysis. Multiple imputation technique will be used to analyze missing data. Every effort will be undertaken to complete any trial participation. Data are recorded by paper Case Report Forms (CRF). For each enrolled study participant a CRF is maintained. The CRFs in this trial are implemented electronically using a dedicated electronic data capturing (EDC) system (REDCap).

Number of Participants with Rationale:

According to the power analysis (power=0.8, one sided Wilcoxon rank sum test, alpha-error 0,05, SD=7, unimportant difference≤3) 69 patients are needed per study arm to state a non-inferiority in both groups. A drop out or lost to follow up rate at approximately 10-15% is expected. Therefore 80 patients are needed per study arm (overall 160 patients).

Statistical Considerations:

Descriptive statistics are used in order to analyse demographic data (age, gender, inability to work, return to work, distribution of occupation, etc.) The main outcome is the OMAS after 12 weeks. The hypothesis is that there is no difference between conservative and surgically treated stable lateral malleolar fractures regarding pain, function, and return to the workplace.

Descriptive statistic with specification of the 95% confidence interval is used for the secondary outcome parameters. If applicable a multivariance analysis is intended.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Acute, stable lateral malleolar fracture

Definition of stable:

* Less than 2mm dislocation in a.p., lateral and gravity-stress x-ray
* Medial tibiotalar distance <4mm and difference <1mm compared to the superior clear space on the gravity-stress and weight bearing x-ray
* No talar subluxation
* No intraoperative instability (Hook-/Frick-Test)

  * Between 18 and 65 years old
  * Living in Switzerland
  * Working
  * Cognitive and physic ability to follow the study protocol

Exclusion Criteria:

* Instable fractures
* Previous ipsilateral surgery on the ankle or foot
* Pregnancy
* Diabetes mellitus
* Neurologic or vascular impairment
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Previous enrolment into the current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Olerud-Molander Ankle Score (OMAS) | after 12 weeks
  The OMAS Score is a patient-reported scale from 0 (totally impaired) to 100 (completely unimpaired) to evaluate subjectively scored function after ankle fracture. It consists of 9 questions: pain (0 to 25), stiffness (0 to 10), swelling (0 to 10), stair climbing (0 to 10), running (0 to 5), jumping (0 to 5), squatting (0 to 5), use of supports (0 to 10), and work/activity level (0 to 20), with higher scores indicating better outcomes

SECONDARY OUTCOMES:
The Visual Analogue Scale Foot and Ankle (VAS FA) | at time of accident, within the first two weeks, after 6 and 12 weeks, after 1, 3 and 5 years
  The VAS FA is a questionnaire based on 20 questions requiring purely subjective answers; 3 different question categories (pain, n=4 questions; function, n=11, other complaints n=5) with a possible maximum of 100 points.
American Orthopedic Foot and Ankle Society Score (AOFAS) | at time of accident, within the first two weeks, after 6 and 12 weeks, after 1, 3 and 5 years
  The AOFAS Score is used for measuring the outcome of treatment in patients who sustained a complex ankle or hindfoot injury. It combines a clinician-reported and a patient-reported part. The questionnaire consists of 9 questions and covers 3 categories: pain (40points), function (50 points) and alignment (10points). These are all scored together for a total of 100 points, indicating no symptoms or impairments.
Foot Function Index (FFI) | at time of accident, within the first two weeks, after 6 and 12 weeks, after 1, 3 and 5 years
  The FFI was developed to measure the impact of foot pathology on function in terms of pain, disability and activity restriction. The FFI questionnaire consists of 18 self-reported items divided into 3 subcategories: pain, disability and activity limitation. The patient has to score each question on a scale from 0 (no pain or difficulty) to 10 (worst pain imaginable or so difficult it requires help). Both total and subcategory scores are calculated.
Return to work | at time of accident, within the first two weeks, after 6 and 12 weeks, after 1, 3 and 5 years
  yes, no or partial (%)
Kellgren-Lawrence scale | at time of accident, within the first two weeks, after 6 and 12 weeks, after 1, 3 and 5 years
  The Kellgren Lawrence grading system is a radiological classification of osteoarthritis. It progresses from grade 0 (no radiographic features of osteoarthritis) to grade IV (signifying severe osteoarthritis) and is based on radiographs.

CONTACTS AND LOCATIONS:
Overall Officials: Fabian Krause, PD Dr., Principal Investigator — Dep. of Orthopaedic Surgery, Inselspital, University of Berne
Locations (1):
- University Hospital Inselspital, BERNE, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided